CLINICAL TRIAL: NCT01688271
Title: A Prospective Study to Determine the Efficacy of Simulation-based Training on Practicing Anesthesiologists' Acquisition of Ultrasound-guided Perineural Catheter Insertion Skills
Brief Title: Simulation-Based Training for Ultrasound-Guided Perineural Catheter Insertion
Status: Completed | Type: Observational
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Edward R. Mariano, Chief, Anesthesiology and Perioperative Care and Associate Professor of Anesthesia Stanford University School of Medicine, VA Palo Alto Health Care System
Other Study IDs: 24882
Record Dates: First submitted 2012-08-29; First posted 2012-09-19 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Pain Management; Simulation; Training; Ultrasonography
Keywords: simulation; ultrasound; perineural infusion; continuous peripheral nerve block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Anesthesiologists

SUMMARY:
This study will determine the efficacy of a teaching program incorporating hybrid simulation in training practicing anesthesiologists on ultrasound (US)-guided continuous peripheral nerve block (CPNB).

This study will also examine the extent of practice change following participation in a regional anesthesia teaching program incorporating hybrid simulation. In addition, this study will assess remaining obstacles to incorporating the use of US-guided perineural catheters through identifying potential future interventions and "tool-kits" for setting up perineural catheter programs.

DETAILED DESCRIPTION:
Study subjects will complete a pre-course survey to assess prior experience then participate in a standardized one-day workshop comprised of two sessions; 1) a didactic lecture and model scanning session and 2) a simulation session. Quantitative and qualitative assessments will be performed using video analysis by two blinded reviewers after equipment orientation (baseline), following first session, and following second session. Performance times, number of attempts, and composite scores for procedural performance and ergonomics will be analyzed within and between groups. Every 3 months for one year, subjects will be surveyed to assess implementation of PNB in practice and identify remaining barriers.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists in practice ten years or more; active board certification (American Board of Anesthesiologists); active license to practice medicine in California; and willingness to spend one full day (8 hours) participating in the standardized workshop and undergo interval survey and interview follow-up for one year.

Exclusion Criteria:

* Formal training (e.g., post-graduate fellowship) in regional anesthesia; current practice includes the routine performance of US-guided PNB (≥10 blocks per month); or visual, hearing, or other communication impairment that would interfere with video recording or require substantial deviation from the standardized teaching curriculum.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active board certificated (American Board of Anesthesiologists) Anesthesiologists in practice ten years or more.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in video assessment score from baseline | baseline (time 0), interval assessment (time 1), and post-course (time 2)
  The primary outcome is the change in composite score from baseline assessment based on the video analysis tool used by blinded reviewers. The baseline assessment at time 0 will take place after initial orientation to the simulation lab. This procedure will take approximately 15 min to perform and record. After the morning session of training (4 hours), the interval assessment at time 1 will take place in the same manner. The final assessment will take place following the entire course (8 hours total) according to the same procedures at time 2. Video recordings will be reviewed at a later date after completion of the training day.

SECONDARY OUTCOMES:
Implementation of new training | Every 3 months post-training for 1 year
  Starting 3 months after the workshop and every 3 months thereafter for one year, subjects will be sent an online practice assessment survey similar to the pre-course survey by the research assistant and will be asked to report their case logs.

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Mariano, MD, MAS, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] Sites BD, Spence BC, Gallagher JD, Wiley CW, Bertrand ML, Blike GT. Characterizing novice behavior associated with learning ultrasound-guided peripheral regional anesthesia. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):107-15. doi: 10.1016/j.rapm.2006.11.006. PMID 17350520
- [Background] Ajmal M, Power S, Smith T, Shorten GD. Ergonomic task analysis of ultrasound-guided femoral nerve block: a pilot study. J Clin Anesth. 2011 Feb;23(1):35-41. doi: 10.1016/j.jclinane.2010.06.006. PMID 21296245
- [Background] Ilfeld BM, Enneking FK. Continuous peripheral nerve blocks at home: a review. Anesth Analg. 2005 Jun;100(6):1822-1833. doi: 10.1213/01.ANE.0000151719.26785.86. PMID 15920221
- [Background] Ilfeld BM, Gearen PF, Enneking FK, Berry LF, Spadoni EH, George SZ, Vandenborne K. Total knee arthroplasty as an overnight-stay procedure using continuous femoral nerve blocks at home: a prospective feasibility study. Anesth Analg. 2006 Jan;102(1):87-90. doi: 10.1213/01.ane.0000189562.86969.9f. PMID 16368810
- [Background] Ilfeld BM, Mariano ER, Williams BA, Woodard JN, Macario A. Hospitalization costs of total knee arthroplasty with a continuous femoral nerve block provided only in the hospital versus on an ambulatory basis: a retrospective, case-control, cost-minimization analysis. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):46-54. doi: 10.1016/j.rapm.2006.10.010. PMID 17196492
- [Background] Sites BD, Chan VW, Neal JM, Weller R, Grau T, Koscielniak-Nielsen ZJ, Ivani G; American Society of Regional Anesthesia and Pain Medicine; European Society Of Regional Anaesthesia and Pain Therapy Joint Committee. The American Society of Regional Anesthesia and Pain Medicine and the European Society Of Regional Anaesthesia and Pain Therapy Joint Committee recommendations for education and training in ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2009 Jan-Feb;34(1):40-6. doi: 10.1097/AAP.0b013e3181926779. PMID 19258987
- [Background] Hadzic A, Vloka JD, Kuroda MM, Koorn R, Birnbach DJ. The practice of peripheral nerve blocks in the United States: a national survey [p2e comments]. Reg Anesth Pain Med. 1998 May-Jun;23(3):241-6. PMID 9613533
- [Background] Kopacz DJ, Neal JM. Regional anesthesia and pain medicine: residency training--the year 2000. Reg Anesth Pain Med. 2002 Jan-Feb;27(1):9-14. doi: 10.1053/rapm.2002.29715. PMID 11799499
- [Background] Kopacz DJ, Neal JM, Pollock JE. The regional anesthesia
- [Background] Marhofer P, Chan VW. Ultrasound-guided regional anesthesia: current concepts and future trends. Anesth Analg. 2007 May;104(5):1265-9, tables of contents. doi: 10.1213/01.ane.0000260614.32794.7b. PMID 17456684
- [Background] Mariano ER, Cheng GS, Choy LP, Loland VJ, Bellars RH, Sandhu NS, Bishop ML, Lee DK, Maldonado RC, Ilfeld BM. Electrical stimulation versus ultrasound guidance for popliteal-sciatic perineural catheter insertion: a randomized controlled trial. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):480-5. doi: 10.1097/AAP.0b013e3181ada57a. PMID 19920423
- [Background] Mariano ER, Loland VJ, Sandhu NS, Bellars RH, Bishop ML, Afra R, Ball ST, Meyer RS, Maldonado RC, Ilfeld BM. Ultrasound guidance versus electrical stimulation for femoral perineural catheter insertion. J Ultrasound Med. 2009 Nov;28(11):1453-60. doi: 10.7863/jum.2009.28.11.1453. PMID 19854959
- [Background] Neal JM, Hsiung RL, Mulroy MF, Halpern BB, Dragnich AD, Slee AE. ASRA checklist improves trainee performance during a simulated episode of local anesthetic systemic toxicity. Reg Anesth Pain Med. 2012 Jan-Feb;37(1):8-15. doi: 10.1097/AAP.0b013e31823d825a. PMID 22157743
- [Background] Boulet JR, Murray DJ. Simulation-based assessment in anesthesiology: requirements for practical implementation. Anesthesiology. 2010 Apr;112(4):1041-52. doi: 10.1097/ALN.0b013e3181cea265. PMID 20234313